CLINICAL TRIAL: NCT00296114
Title: Pancreatic Cancer Serum and DNA Repository
Status: Completed | Type: Observational
Sponsor: Pancreatic Cancer Research Team (Other)
Responsible Party: Sponsor
Other Study IDs: PCRT 03 001; NCT00250107 (obsolete NCT alias)
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2011-12

CONDITIONS: Pancreas Cancer
Keywords: Cancer; Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood and Serum Samples

INTERVENTIONS:
Procedure: Serum and DNA Samples — To collect serum and DNA samples from subjects

SUMMARY:
To prospectively collect serum and DNA samples from subjects with pancreatic cancer, pancreatitis, liver disease, and from healthy and at-risk volunteers in order to identify novel biomarkers for early diagnosis, differential diagnosis, stage, natural history of the disease, response to treatment, and to identify novel targets for therapeutic interventions. In particular:

DETAILED DESCRIPTION:
* To establish a central pancreatic cancer specimen repository to serve as a resource for current and future scientific studies.
* To utilize the PCRT clinical data base to perform clinicopathologic correlation with the results of those studies.
* To test new hypotheses as they emerge.

ELIGIBILITY:
Inclusion Criteria:

Ages Eligible for Study: 18 Years and above, Genders Eligible for Study: Both

Criteria

Inclusion Criteria:

4.1 At the time of subject registration, CRAB will verify the institution's IRB date to ensure that the subject can be enrolled.

4.2 Potential study participants must meet the eligibility criteria found in Section 12.0 (Eligibility Checklist). Candidates will fall into one of four groups:

1. Pancreatic cancer patients;
2. Pancreatic and Liver Disease patients;
3. Healthy, At-Risk Volunteers (smoker, (defined as individuals who have smoked >= 100 cigarettes in their lifetime, and who currently smoke every day or some days [MMWR November 12, 2004, 53(44);1035-1037]), diabetic, and/or family history); and
4. Healthy Volunteers (no history of cancer). The Eligibility Checklist must be photocopied, completed and stored on site. Eligibility is confirmed during registration, by answering yes to the question, Have all eligibility criteria been met? on the Registration Form.

Eligibility Checklist:

1. Pancreatic Cancer Patient Criteria All subjects, regardless of gender and ethnicity are eligible for this study Pathological diagnosis of pancreatic malignant neoplasm Expected availability of clinical follow up data Eighteen years old or older All subjects must be informed of the investigational nature of this protocol Written, informed consent obtained in accordance with institutional and federal guidelines
2. Pancreatitis and Liver Disease Subject Criteria All subjects, regardless of gender and ethnicity are eligible for this study Pathological diagnosis of pancreatitis or liver disease Eighteen years old or older All subjects must be informed of the investigational nature of this protocol Written, informed consent obtained in accordance with institutional and federal guidelines
3. Healthy, At-Risk Volunteers All subjects, regardless of gender and ethnicity are eligible for this study Is a smoker, is diabetic AND/OR has a family history of pancreatic cancer Eighteen years old or older with no history of cancer All subjects must be informed of the investigational nature of this protocol Written, informed consent obtained in accordance with institutional and federal guidelines
4. Healthy Volunteers (no at-risk factors) All subjects, regardless of gender and ethnicity are eligible for this study Eighteen years old or older with no history of cancer All subjects must be informed of the investigational nature of this protocol Written, informed consent obtained in accordance with institutional and federal guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Samples are collected on: Pancreatic Cancer, Liver Disease, Pancreatitis, Healthy and Healthy at Risk Subjects.
Sampling Method: Non-Probability Sample
Enrollment: 690 (Actual)
Dates: Start 2004-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, MD, PhD, Study Chair — Hospital Universitario Sanchinarro, Madrid, Spain
Locations (10):
- United States (9):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - University of Arizona/Arizona Cancer Center, Tucson, Arizona
  - UCLA Medical Center, Los Angeles, California
  - RUSH University Medical Center, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center/Johns Hopkins, Baltimore, Maryland
  - Abbott Northwestern Hospital/Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - University of New Mexico, Albuquerque, New Mexico
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - South Texas Oncology and Hematology, San Antonio, Texas
- University Hospital (12 De Octubre), Madrid, Spain

REFERENCES:
- See also: Pancreatic Cancer Research Team - Public/Members — http://www.pcrt.org/